CLINICAL TRIAL: NCT03680625
Title: Virtual Reality Compared to Passive Distraction for Pain Management During Orthopedic Procedures in Children: A Randomized Controlled Trial.
Brief Title: Virtual Reality vs Passive Distraction for Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Montreal Children's Hospital of the MUHC (Other); Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-2030
Record Dates: First submitted 2018-07-10; First posted 2018-09-21 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Virtual Reality; Pain; Pain Perception; Pain Management; Anxiety; Catastrophizing, Pain; Stress
Keywords: Virtual reality; Immersive distraction; Virtual world; Virtual environment; Passive distraction; Procedural pain; Procedural anxiety; Acute pain; Pain management; Anxiety; Children, Child; Kid, Kids; Pediatric, Pediatrics; Young children; Orthopedics; Kirschner wire, K pin; Bone wires; Percutaneous pins; Non-pharmacological; Clinical Research; Nursing Practice; User-computer interface; Pediatric Nursing; Hospital, Pediatric; Sutures; Stress
MeSH Terms: conditions — Pain; Agnosia; Anxiety Disorders; Pain, Procedural; Acute Pain; Deafness, Autosomal Recessive 1A

STUDY DESIGN:
Intervention Model Description: parallel/2 groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive Distraction (Active Comparator): The child will watch a video on an iPad® during the pin removal procedure and/or removal of sutures.
  Interventions: Device: Passive Distraction
- Virtual Reality Distraction (Experimental): The child will visualize and interact with the virtual environment using an Oculus Quest® head-mounted device throughout the pin removal procedure and/or removal of sutures.
  Interventions: Device: Virtual Reality Distraction

INTERVENTIONS:
Device: Passive Distraction — Patients in this group will be offered an iPad® showing a video while they will undergo their pins' removal and/or removal of sutures. There will be videos appropriate for each age group. The child can choose from the videos presented on the iPad® and start watching 5 minutes before the beginning of the procedure to assure similar preparation for both groups.
  Arms: Passive Distraction
Device: Virtual Reality Distraction — Patients in this group will be offered virtual reality distraction through the use of Oculus Quest® while they undergo their pins' removal and/or removal of sutures. VR produces a high level of immersion, with high photorealism while maintaining the low latency necessary to induce presence and prevent cybersickness symptoms such as nausea, vomiting, headache. The videogame was developed by our team with three levels of difficulty, and approved by pediatric healthcare professionals. The game, oculus head-mounted device and computer will be available in the procedure room and ready for immediate use. The head-mounted device will be adjusted to the head of the child before any procedure and a period of 5 minutes will be allotted prior to pin and/or suture removal in order for the child to get acquainted with the game and immersed in the virtual environment.
  Arms: Virtual Reality Distraction

SUMMARY:
Background: Outpatient pediatric orthopedic procedures such as percutaneous pins removal and sutures are considered painful and generate significant stress and anxiety in children. However, given their short duration and the need for a quick turnover in outpatient clinics, there are very few interventions aimed at relieving pain, stress and anxiety related to these procedures. Neither simple analgesia nor topical anesthetics proved effective for procedural pain reduction with this population. Moreover, narcotics and procedural sedation do not appear to be feasible alternatives as they require surveillance, prolonging visit to the outpatient clinic and generating several undesired side effects. Therefore, it would be imperative to explore non-pharmacological pain management methods as they require minimal preparation and do not usually generate any side effects.

Aim: To examine the effect of virtual reality (VR) compared to passive distraction, on pain, stress, anxiety and memory of pain in children undergoing a percutaneous pin removal procedure or sutures in an outpatient orthopedic clinic.

Hypothesis: VR distraction provides better pain relief during percutaneous pin removal procedures or sutures than passive distraction, in children from 7 to 21 years old.

Methods: The study will be a prospective randomized controlled trial with parallel groups. Children from 7 to 21 years old, visiting the clinic for follow up and percutaneous pin removal procedure or sutures, accompanied by a parent or legal guardian will be recruited. The experimental group will receive a VR distraction through a head-mounted Oculus Quest® and the control group will receive passive distraction through watching a video on an iPad®. The primary outcome will be the mean pain score after the procedure (self-report of pain level during the procedure) measured by the Numerical Rating Scale (NRS). Anxiety will be measured by the Child Fear Scale (CFS) and stress will be measured using level of salivary Alpha-Amylase before and 10-min after the procedure. Memories of pain and anxiety will be measured one week after the procedure using the same scales (NRS and CFS). The investigators aim to recruit 188 children.

Discussion: The investigators believe that results of this study will allow to improve pain, stress and anxiety management practices in this orthopedic clinic by showing that non-pharmacological interventions can be done, at very low cost, to improve the experience of the child undergoing these painful procedures through an innovative and more humanistic approach.

DETAILED DESCRIPTION:
BACKGROUND

In children, many fractures treated surgically will be stabilized percutaneously with Kirschner wires and some will require sutures to help the surgical wound to heal. When the fracture is adequately healed, the percutaneous wires and/or the sutures are generally removed in the outpatient clinic. These procedures represent a potential source of pain, stress and anxiety for the patient, as well as for the parents and the caregivers.

A study looked at different types of analgesia during percutaneous pin removal comparing Acetaminophen, Ibuprofen and placebo but no clinically nor statistically significant difference was found among the three groups. Another study compared topical liposomal lidocaine to a placebo but found no statistically significant difference in postprocedure pain scores between groups. On the other hand, administration of narcotics or procedural sedation for pin removal procedure probably exceeds the real needs for the majority of patients. Adding the fact that the administration of narcotics or procedural sedation requires monitoring post administration, those options lengthen visit time, reduce significantly the efficiency in an outpatient clinic setting and are not recommended for routine administration.

In contrast, there seems to be some emerging evidence about distraction methods such as distraction techniques facilitated by a hospital play specialist for pin removal procedures. Distraction use for children in orthopedic outpatient clinics has been reported anecdotally in some literature but, to our knowledge, has never been formally assessed in a randomised controlled trial. Exploring non-pharmacological interventions, including distraction, could be a promising venue for pain management in this population as they are simple, practical, easily implementable and usually without side effects.

Virtual Reality (VR) is a distraction method that allows the user to interact with an immersive environment generated by a computer stimulating different senses. A review of studies on VR, mostly conducted with adult burn patients, showed a 35 to 50% reduction in procedural pain while using VR. Its positive effect has also been reported on anxiety and general distress during painful medical procedures in children and in adults such as venipuncture, wound care, chemotherapy, dental procedures, etc. A recent randomized-controlled trial comparing VR and standard distraction in children undergoing blood drawn procedures, demonstrated a significant positive effect of VR on pain and anxiety reduction as well as patients', caregivers' and phlebotomist's satisfaction. The authors also concluded that VR was more effective for children with higher anxiety sensitivity, adding another plus value to this new technology in children's care.

There is evidence to suggest that reducing procedural pain and distress in the short-term, will have long lasting effects on children's pain and health trajectories in the long-term. The effect of pain on a developing child does not end after painful procedures end; how children remember these experiences can have long lasting effects. Children who recall pain in negatively-biased ways experience more pain and distress at future pain experiences and are at risk for developing persistent pain problems and fears and avoidance of medical care. Importantly, children (and parents) who are more anxious and distressed prior to painful medical procedures, and who experience higher pain during medical procedures, are the very children who develop these negatively biased recalls. Therefore, we will also examine the effect of VR distraction, a more immersive intervention, on children's later recall of pain. This is innovative as we did not find any other studies using VR and collecting data on pain and anxiety recalls in children following painful medical procedures. Further, we will compare salivary Alpha-Amylase levels between groups, which is a reliable and valid surrogate marker of stress that increases in response to physical and psychological stressful conditions such as experience of medical procedures.

Considering the lack of optimal pain, stress and anxiety management during pin removal and/or removal or sutures, and the positive effect of VR for painful procedures, combining VR to pin/sutures removal procedures may show promising results. To our knowledge, no other studies have tested the effect of VR distraction via Oculus Quest® for procedural pain management in children undergoing painful orthopedic procedures such as percutaneous pins removal and removal of sutures.

AIM & STUDY OBJECTIVES

Primary objective: To determine if VR distraction provides better pain relief during percutaneous pin removal procedures and/or removal of sutures, than passive distraction, in children from 7 to 21 years old.

Secondary Objectives:

1. To determine if VR distraction provides better anxiety and stress relief in children during percutaneous pin removal procedures and/or removal of sutures than passive distraction.
2. To determine if children receiving VR distraction will remember less pain and anxiety than children receiving passive distraction during the percutaneous pin removal procedure and/or removal of sutures.
3. To compare the occurrence of side effects between VR distraction and passive distraction groups.
4. To compare healthcare professionals' satisfaction levels between VR distraction and passive distraction.
5. To compare children and parents' satisfaction levels between VR distraction and passive distraction.
6. To compare requirement for rescue analgesia between VR distraction and passive distraction.
7. To compare mean levels of physiological stress between groups (Levels of salivary Alpha-Amylase - Surrogate marker of stress)

METHODS

Design: Multi-center randomized controlled trial using a parallel design with two groups: a) experimental group (virtual reality), b) active comparator (videogame on an iPad®).

Sample and Setting: Recruitment will be done through convenience sampling at the orthopedic outpatient day clinic at CHU Ste-Justine, and at the Shriners Hospital for Children and the Montreal Children's Hospital.

Measures and outcomes: Timepoints. Data will be collected by the research assistant at the following study times: before the procedure to establish baseline (T0), immediately after the procedure (T1), and one week after the procedure (T2).

Sample Size: Group sample sizes of 94 and 94 (188 in total) are necessary to achieve 80% power to reject the null hypothesis of equal means when the population mean difference for pain is 1.5 with a standard deviation for both groups of 3.3 and a significance level (alpha) of 2.5% using a two-sided t-test. Group sample sizes of 67 and 67 (134 in total) are necessary to achieve 80% power to reject the null hypothesis of equal means when the population mean difference for anxiety is 0.7 with a standard deviation for both groups of 1.3 and a significance level (alpha) of 2.5% using a two- sided t-test. Based on our pilot's study data, there were no attrition. No interim analysis will be conducted.

Data analysis plan: Descriptive statistics will be used to present sociodemographic and clinical data as well as parents, children and healthcare professionals' levels of satisfaction. Primary analyses: An ANCOVA adjusted for centers and baseline (T0) pain score measurement/anxiety score measurement will be used to assess the mean difference in pain scores on the NRS scale/the mean difference in anxiety scores on the CFS, between the experimental and the control groups at T1. Analyses will be carried out according to the intention-to-treat principle, with a significance level (α) of 0.025. Secondary analyses: Secondary analyses using ANCOVA adjusted for centers and pain score measurement/anxiety score measurement at T1 will be used to assess the mean difference in pain memories/anxiety memory between the experimental and the control groups at T2. An ANOVA adjusted for centers will be used to assess mean differences in children-reported pain on the GRS between the experimental and the control groups at T1. Correlations will be calculated to compare stress level between groups. Cochran-Mantel-Haenszel tests will be conducted to compare dichotomous variables including the occurrence of side effects, use of rescue analgesia, and use of other non-pharmacological interventions in each group.

ELIGIBILITY:
Inclusion Criteria:

* Requiring a percutaneous pins and/or sutures removal procedure,
* Accompanied by a consenting parent or legal guardian who can understand, read and write either French or English.

Exclusion Criteria:

* Having a diagnosed cognitive impairment preventing them from interacting with the games or answering questions related to pain, anxiety, and pain memory,
* Have a diagnosis of epilepsy or any other condition precluding them from playing a virtual reality game,
* Cannot be in a sitting or semi-upright sitting position (Fowler's position) during the procedure as the game in the virtual reality group requires an angle of at least 45 degrees for head-tracking.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Pain intensity | T1, immediately after the procedure.
  self-report of pain level during the procedure assessed using the Numerical Rating Scale (NRS) ranging from 0 to 10; 0=no pain to 10=pain as bad as it could be.
Anxiety level | T0, before the procedure (baseline); T1, immediately after the procedure.
  Children's Fear Scale (CFS)(0-4)

SECONDARY OUTCOMES:
Presence in the game | T1, immediately after the procedure
  Graphic Rating Scale (GRS) consisting of seven items to measure the cognitive, the affective and the sensory components related to presence in the game and pain on a scale of 0 to 10.
Stress | T0, before the procedure (baseline); T1, immediately after the procedure.
  Salivary mouth swab for measurement of Alpha-Amylase
Parents' and children's satisfaction levels | T1, immediately after the procedure
  0 to 10 numerical scale
Healthcare professionals' satisfaction level | An average of one year after the beginning of the study (mid-recruitement)
  tailored questionnaire with four choices response scale from Strongly agree to Strongly disagree for 7 items related to their level of satisfaction with the intervention and its effect on the procedure.
Analgesic requirement | T1, immediately after the procedure
  Need for rescue medication administered during the pin removal procedure (yes/no).
Co-interventions | T1, immediately after the procedure
  Use of other non-pharmacological interventions (parental distraction, music/singing, comforting, or other) during the procedure. (yes/no)
Side effects | T1, immediately after the procedure.
  Occurrence of side effects during or after the procedure related to the research interventions.
Children's memory of pain | T2, one week after the procedure
  The same Numerical Rating Scale (NRS) (0-10) administered during the initial session to measure pain but framed in terms of recall.
Children's memory of anxiety | T2, one week after the procedure
  The same measure Children's Fear Scale (CFS) (0-4) administered during the initial session to measure anxiety but framed in terms of recall.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, PhD, Principal Investigator — St. Justine's Hospital
Locations (3):
- Canada (3):
  - St. Justine's Hospital, Montreal, Quebec
  - Shriners Hospitals for Children, Montreal, Quebec
  - Montreal Children's Hospital of the MUHC, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guingo E, Debeurme MH, Dos Santos RP, Addab S, Rainville P, Bouchard S, Chougui K, Tsimicalis A, Nault ML, Ducruet T, Ledjiar O, Noel M, St-Arneault K, Cotes-Turpin C, Hung N, Ouimet P, Parent S, Gardner J, Bernstein M, Le May S. Efficacy of Virtual Reality vs. Tablet Games for Pain and Anxiety in Children Undergoing Bone Pins Removal: Randomised Clinical Trial. J Adv Nurs. 2026 Feb;82(2):1791-1802. doi: 10.1111/jan.16991. Epub 2025 Apr 29. PMID 40302143
- [Derived] Le May S, Tsimicalis A, Noel M, Rainville P, Khadra C, Ballard A, Guingo E, Cotes-Turpin C, Addab S, Chougui K, Francoeur M, Hung N, Bernstein M, Bouchard S, Parent S, Hupin Debeurme M. Immersive virtual reality vs. non-immersive distraction for pain management of children during bone pins and sutures removal: A randomized clinical trial protocol. J Adv Nurs. 2021 Jan;77(1):439-447. doi: 10.1111/jan.14607. Epub 2020 Oct 24. PMID 33098330